CLINICAL TRIAL: NCT05388773
Title: Phase II Trial of Transoral Surgical Resection Followed by De-escalated Adjuvant IMRT in Resectable p16+ Locally Advanced Oropharynx Cancer
Brief Title: Transoral Surgical Resection Followed by De-escalated Adjuvant IMRT in Resectable p16+ Locally Advanced Oropharynx Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Heath Skinner (Other)
Responsible Party: Sponsor-Investigator, Heath Skinner, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-030
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Oropharynx Cancer
Keywords: Papillomavirus Infections; Carcinoma, Squamous Cell; Oropharyngeal Neoplasms; Papilloma; Neoplasms, Glandular and Epithelial; Pharyngeal Neoplasms; Otorhinolaryngologic Neoplasms; Head and Neck Neoplasms; Pharyngeal Diseases; Stomatognathic Diseases; Otorhinolaryngologic Diseases; DNA Virus Infections; Tumor Virus Infections; Antineoplastic Agents; Intensity Modulated Radiotherapy; Carboplatin; Cisplatin; Transoral Surgery
MeSH Terms: conditions — Oropharyngeal Neoplasms; Papillomavirus Infections; Carcinoma, Squamous Cell; Papilloma; Neoplasms, Glandular and Epithelial; Pharyngeal Neoplasms; Otorhinolaryngologic Neoplasms; Head and Neck Neoplasms; Pharyngeal Diseases; Stomatognathic Diseases; Otorhinolaryngologic Diseases; DNA Virus Infections; Tumor Virus Infections | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm S (Low Risk) (Experimental): Low risk patients are defined as T1-T2 AND 0 or 1 metastatic lymph nodes AND <3 cm AND clear (≥3mm) margins AND no extracapsular extension (ECE) AND no perineural invasion AND no lymphovascular invasion.
  Patients will undergo transoral surgical resection of the oropharyngeal tumor.
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: quality-of-life assessment
- Arm RT (Intermediate Risk) (Experimental): Intermediate risk patients are defined as having any of the following features: One or more close (<3mm) margins, OR "minimal" ≤1 mm ECE OR 1 or more metastatic lymph nodes >3 cm in diameter OR 2-4 lymph nodes positive (≤ 6 cm in diameter), OR perineural invasion OR lymphovascular invasion
  Patients will undergo transoral surgical resection of the oropharyngeal tumor. Following surgery, patients will receive low-dose IMRT five times a week for 3 weeks.
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: quality-of-life assessment; Radiation: intensity-modulated radiation therapy
- Arm CRT (High Risk) (Experimental): High risk patients are defined as having any of the following features: One or more positive margins OR >1 mm ECE OR ≥ 5 metastatic lymph nodes.
  Patients will undergo transoral surgical resection of the oropharyngeal tumor. Following surgery, patients will receive low-dose IMRT six times a week and a weekly chemotherapy infusion (cisplatin or carboplatin) during radiation therapy.
  Patients will receive 2 Gy/fraction, 6 fractions per week with at least a 6-hour interfraction interval between each treatment:
  * PTV-P50 or PTV-N50: 50 Gy in 25 fractions (2 Gy/fx)
  * PTV-N45: 45 Gy in 25 fractions (1.8 Gy/fx) with simultaneous integrated boost to the PTV-P50 volume.
  * PTV-P30 or PTV-N30: 30 Gy in 15 fractions (2 Gy/fx)
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: quality-of-life assessment; Radiation: intensity-modulated radiation therapy; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Transoral surgical resection of tumor(s).
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies.
  Other Names: quality of life assessment
Radiation: intensity-modulated radiation therapy — Low-dose IMRT
  Other Names: IMRT
  Arms: Arm CRT (High Risk); Arm RT (Intermediate Risk)
Drug: Cisplatin — Given IV.
  Other Names: CACP; CDDP; CPDD; DDP
  Arms: Arm CRT (High Risk)
Drug: Carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Arm CRT (High Risk)

SUMMARY:
This is a trial studying patients with human papilloma virus (HPV) positive oropharyngeal cancer with tumors that can be removed via transoral surgery. Following surgery, patients will be classified as either low, intermediate, or high risk based on the characteristics of the tumors. Low risk patients (Arm S) will receive no further treatment after surgery. Intermediate risk patients (Arm RT) will be treated with Intensity Modulated Radiotherapy (IMRT) after surgery. High risk patients (Arm CRT) will receive a combination of IMRT and chemotherapy after surgery. Patients will be followed for up to five years after the completion of treatment.

DETAILED DESCRIPTION:
This phase II trial is designed to rationally de-escalate adjuvant (Intensity Modulated Radiotherapy (IMRT) in the post-transoral surgery (TOS) setting in a study population consisting of patients with resectable oropharynx carcinoma, p16+ as confirmed by immunohistochemistry IHC, with a performance status (PS) of 0-1. Patients will be classified into one of three category/treatment groups (low-, intermediate-, and high-risk) according to their highest pathologically risk feature. Radiation will be given via an IMRT technique. For the high-risk patient group, a reduced, but slightly accelerated radiotherapy (RT) fractionation regimen of 50 Gy (HCC 18-034) in conjunction with cisplatin will be used compared to the standard 66 Gy and cisplatin. Low risk patients will transition to observation, intermediate risk patients will receive 30 Gy in 15 fractions of IMRT, and high risk patients will receive 50 Gy in 25 fractions (one day a week will include two treatments) plus 40 mg/m2 Cisplatin for 5 weeks. Patients who are not able to tolerate cisplatin will receive carboplatin instead.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1 or Karnofsky score 80-100.
* Preference is to register patients prior to surgery. However, if not registered prior to surgery, the patient can be registered prior to adjuvant therapy.
* Patients must have newly diagnosed, histologically or cytologically confirmed SCC or undifferentiated carcinoma of the oropharynx. Patients must have been determined to have resectable oropharyngeal disease. Patients with primary tumor or nodal metastasis fixed to the carotid artery, skull base or cervical spine are not eligible.
* Patients must be deemed eligible for a TOS procedure with no evidence of distant metastasis as determined by imaging studies. Metastatic disease may be evaluated using CT or PET/CT where appropriate; this can be performed with or without contrast. The following imaging is acceptable to evaluate the primary and regional disease:

  * CT Neck (with contrast preferred but not required)
  * PET/CT
  * MRI Neck (contrast preferred but not required)
* Patients must have biopsy-proven p16+ oropharynx cancer; the histologic evidence of invasive squamous cell carcinoma may have been obtained from the primary tumor or metastatic lymph node. It is required that patients have a positive p16 IHC (as surrogate for HPV) status from either the primary tumor or metastatic lymph node.
* Carcinoma of the oropharynx associated with HPV as determined by p16 protein expression using immunohistochemistry (IHC) performed by a CLIA approved laboratory. Using p16 antibody obtained from Roche mtm laboratories AG (CINtec, clone E6H4) is recommended.
* No prior radiation above the clavicles.
* Patients with a history of a curatively treated malignancy must be disease-free for at least two years except for carcinoma in situ of cervix, melanoma in-situ (if fully resected), and/or non- melanomatous skin cancer.
* Patients with the following within the last 6 months prior to registration must be evaluated by a cardiologist and/or neurologist prior to entry into the study.

  * Congestive heart failure > NYHA Class II
  * CVA/TIA
  * Unstable angina
  * Myocardial infarction (with or without ST elevation)
* Patients must have acceptable renal and hepatic function within 4 weeks prior to registration

  o For patients stratified following surgery and to concurrent chemotherapy (Arm CRT), calculated creatinine clearance must be > 60 ml/min using the Cockcroft-Gault formula
* In patients with a contraindication to cisplatin, carboplatin can be used at time of patient enrollment if they are allocated to ARM CRT.

Exclusion Criteria:

* No evidence of extensive or "matted/fixed" pathologic adenopathy on preoperative imaging.
* Patients must not need a microvascular (free flap) reconstruction. Women must not be pregnant or breast-feeding due to the teratogenicity of chemotherapy. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Patient must not have an intercurrent illness likely to interfere with protocol therapy or prevent surgical resection
* Patients must not have uncontrolled diabetes, uncontrolled infection despite antibiotics, or uncontrolled hypertension within 30 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 2 years (for cohort)
  Time to recurrence, defined as local and/or regional progression (identification of disease growth that is present within the area in which it was first located) and/or distant metastasis (identification of disease growth that is present in area(s) distant to that previously located). Local progression is defined as progression at the primary tumor site. Regional progression is defined as progression in the draining lymphatics (typically the cervical, retropharyngeal/retrostyloid and supraclavicular lymph nodes). Distant progression is defined as tumor recurrence in one or more non-local and non-regional sites (e.g., bone, lung, liver, etc.). Recurrent malignancy will be determined based on clinical exam and imaging findings. Patients who are disease-free but who die from other causes will be censored.

SECONDARY OUTCOMES:
Loco-regional control (at 1 year) | Up to 1 year
  Loco-regional control will be evaluated based on the percentage of patients without recurrence (identification of disease growth) in the primary site or regional lymphatics based on imaging and/or clinical exam.
Loco-regional control (at 2 years) | Up to 2 year
  Loco-regional control will be evaluated based on the percentage of patients without recurrence (identification of disease growth) in the primary site or regional lymphatics based on imaging and/or clinical exam.
Time to distant metastasis (at 1 year) | Up to 1 year
  Percentage of patients with distant metastasis (identification of disease growth that is present in area(s) distant to that previously located) evident on imaging and/or clinical exam. Distant metastasis is defined as tumor recurrence in one or more non-local (at the primary tumor) and non-regional (draining lymphatic) sites such as bone, lung, liver, etc.
Time to distant metastasis (at 2 years) | Up to 2 years
  Percentage of patients with distant metastasis (identification of disease growth that is present in area(s) distant to that previously located) evident on imaging and/or clinical exam. Distant metastasis is defined as tumor recurrence in one or more non-local (at the primary tumor) and non-regional (draining lymphatic) sites such as bone, lung, liver, etc.
Overall survival at 1 year | Up to 1 year
  Overall survival will be measured as the time from start of treatment to death from any cause.
Overall survival at 2 years | Up to 2 years
  Overall survival will be measured as the time from start of treatment to death from any cause.
Distribution of patients based on histologic risk features | Up to 3 years
  The percentage of total patients enrolled in the study allocated to low (Arm S), intermediate (Arm RT) and high risk (Arm CRT) groups. Histologic risk features are defined as follows: Low risk (ARM S) - T1-T2 AND 0 or 1 metastatic lymph nodes AND <3 cm AND clear (≥3mm) margins AND no extracapsular extension (ECE) AND no perineural invasion AND no lymphovascular invasion; Intermediate risk (ARM RT) - Any of the following features: One or more close (<3mm) margins, OR "minimal" ≤1 mm ECE OR 1 or more metastatic lymph nodes >3 cm in diameter OR 2-4 lymph nodes positive (≤ 6 cm in diameter), OR perineural invasion OR lymphovascular invasion; High risk (ARM CRT) - Any of the following features: One or more positive margins OR >1 mm ECE OR ≥ 5 metastatic lymph nodes.
Assessment of PEG tube dependence | At 1 year (post treatment)
  The percentage of patients that have a feeding tube, by Arm, for the low (Arm S), intermediate (Arm RT) and high risk (Arm CRT) groups following treatment with transoral resection and adjuvant therapy.
Adverse Events Related to Treatment | Up to 5 years
  Number of patients experiencing toxicities related to study treatment per Common Terminology Criteria for Adverse Events (CTCAE v5.0) determined at each follow-up summarized by frequency and grade.
Quality of Life via FACT-HN | Baseline (before treatment), at 4-8 weeks post-surgery, at 3 months, 6 months, 1 year, up to 2 years following treatment
  FACT-HN is a self-administered questionnaire. Item responses are on a Likert scale score ranging from 0 to 4. Individual responses are summed to compute subscale scores, and the subscales to compute overall total scores. FACT-HN includes 2 parts - FACT-G and FACT-HN. The basic FACT-G (general) is comprised of 27 items, with four subscales including Physical Well-Being (score = 0-28), Social/Family Well-Being (score= 0-28), Emotional Well-Being (score = 0-24), and Functional Well-Being, (score = 0-28), for a total score min/max = 0-108. The FACT-HN is comprised of 12 head and neck specific items (0-48). Thus, the overall total possible score range is 0-156. Analysis will include the FACT Head & Neck Trial Outcome Index, a composite score which includes only physical, functional, and FACT-HN, thus, scores range from 0-104. Higher scores indicate better Quality of Life.
MD Anderson Symptom Inventory-Head & Neck (MDASI-HN) | Baseline (before treatment), at 4-8 weeks post-surgery, at 3 months, 6 months, up to 2 years following treatment
  Patient-reported swallowing perception and performance using MDASI-HN measures treatment related symptom burden in head and neck cancer patients. The 20-item MDASI measures both severity and burden of symptoms and their effect on patients' daily activities, using a numeric rating scale of 0-10. This instrument includes 13 core symptoms and 9 head and neck specific items. Higher scores indicate superior perception of function.
Modified Barium Swallow (MBS) rating | Before treatment, at 4-8 weeks post-surgery, 6 months and 24 months following treatment
  Three swallowing outcomes will be rated by the SLP conducting the MBS study and reported by research staff: 1) laryngeal penetration (yes, no); 2) aspiration (no, sensate, silent), and 3) pharyngeal residue (no, < 50%, > 50%). These have been selected as universal items generally reported by swallowing clinicians that have been shown to significantly predict pneumonia in patients with oropharyngeal cancers. Prevalence of these dysphagia endpoints will be estimated at each time point.
Voice outcomes | Baseline (before treatment), at 4-8 weeks post-surgery, at 1 year, up to 2 years following treatment
  Patient-reported voice outcomes will be assessed using the Voice Handicap Index-10 (VHI-10) survey. The VHI-10 is a patient self-assessment instrument that quantifies patients' perception of their voice handicap. It evaluates patient's physical (P), emotional (E), and functional (F) perceptions of voice and has shown to be highly reliable for internal consistency and test-retest stability. The VHI-10 utilizes a 10-item questionnaire in which the patient circles the response that most accurately reflects his or her own experience on a linear scale (from "never" to "always"). "Always" response is scored 4 points, a "Never" response is scored 0. The remaining options are scored between 1 and 3 points. The tallied number of points for each of the subscales is computed to a total composite score. The patient's values are compared to published norms.
Performance Status Scale (PSS-HN) | Baseline (before treatment), at 4-8 weeks post-surgery, at 3 months, 6 months, 1 year, up to 2 years following treatment
  The Performance Status Scale (PSS-HN) is a clinician-rated instrument consisting of 3 questions: normalcy of diet, public eating/swallowing, and understandability of speech subscales in patients with head and neck cancer. Each subscale is rated from 0 to 100, with higher scores indicating better performance.
MD Anderson Dysphagia Inventory (MDADI) | Baseline (before treatment), at 4-8 weeks post-surgery, at 1 year, up to 2 years following treatment
  Patient-reported swallowing-related quality of life will be measured using the MD Anderson Dysphagia Inventory (MDADI). It evaluates the patient's physical (P), emotional (E) and functional (F) perceptions of swallowing dysfunction. The MDADI is a 20-item questionnaire in which the patient circles the response that best reflects their experience in the past week on a 5-point Likert Scale with answers ranging from "Strongly Agree" (scored as 1 point on all questions except E7 and F2, where it is scored as 5 points) to "Strongly Disagree" (scored as 5 points on all questions except E7 and F2, where it is scored as 1 point). Scores for individual questions are summed and averaged to obtain a composite score ranging from 20 (extremely low swallow functioning) to 100 (high swallow functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Heath Skinner, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No